CLINICAL TRIAL: NCT04901273
Title: Homologous PRP Versus Placebo in the Infiltrative Treatment of Knee Osteoarthritis in Over 65 Years Old Patients.
Brief Title: Homologous PRP vs Placebo in Knee Osteoarthritis in Over 65 Years Old Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRP-o65
Record Dates: First submitted 2021-05-17; First posted 2021-05-25 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis
Keywords: knee; knee osteoarthritis; PRP; Homologous PRP; PRP injections; injection treatment; Randomized controlled trial; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: The study is a double-blinded RCT with possibility ,after 6 months, to cross-over from control arm (saline solution ) to the treatment arm (Homologous PRP). After 6 months, patients in the control arm have the possibility to cross-over into the treatment arm, in which case they will be followed for an additional 12 months.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind randomized controlled trial with 1:1 allocation. Patient blinding will be provided during the injection treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Homologous PRP (Experimental): This group of patients will be treated with single intra-articular injection of Homologous PRP. At the 6-month follow-up visit, the patient will be informed about the treatment received.
  Interventions: Procedure: Homologous PRP injections
- Saline solution (Placebo Comparator): This group of patients will be treated with single intra-articular injection of saline solution (placebo). At the 6-month follow-up visit, patients will be informed about the treatment received. Patients of this group can cross-over to the treatment arm after 6 months.
  Interventions: Procedure: Placebo injection (saline solution)

INTERVENTIONS:
Procedure: Homologous PRP injections — Patients will be treated with a single injection of Homologous PRP (5 ml) in the knee joint affected by osteoarthritis.
  Arms: Homologous PRP
Procedure: Placebo injection (saline solution) — Patients will be treated with a single injections of saline solution (5 ml) in the knee joint affected by osteoarthritis
  Arms: Saline solution

SUMMARY:
The aim of the study is to compare the 6 months clinical outcome of the treatment with a single injection of Homologous PRP versus single injection of placebo (saline solution) in the infiltrative treatment of knee osteoarthritis in over 65 years old patients. The evaluation will be performed through clinical, subjective and objective assessments.

DETAILED DESCRIPTION:
204 patients affected by knee osteoarthritis will be included in a double-blinded RCT with possibility ,after 6 months, to cross-over from control arm ( saline solution ) to the treatment arm (Homologous PRP). Patients will be followed-up with clinical evaluation at 1,3 and 6 months. During the follow-up visits ,will be evaluated the inflammatory status of the knee by thermographic assessment. Patients in the treatment arm (Homologous PRP) will be followed for an additional 6 months (up to 12 months of follow-up). After 6 months, patients in the control arm have the possibility to cross-over into the treatment arm, in which case they will be followed for an additional 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral involvement;
2. Signs and symptoms of degenerative pathology of the knee cartilage;
3. Radiographic or MRI signs of degenerative pathology of the knee cartilage (Kellgren-Lawrence 1-4 grades);
4. Ability and consent of patients to actively participate in clinical follow-up;
5. Signature of informed consent

Exclusion Criteria:

1. Patients undergoing knee surgery within the previous 12 months;
2. Patients with malignant neoplasms;
3. Patients with rheumatic diseases;
4. Patients with diabetes;
5. Patients with hematologic diseases (coagulopathies);
6. Patients with metabolic disorders of the thyroid gland;
7. Patients abusing alcoholic beverages, drugs or medications
8. Body Mass Index > 35

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
KOOS-Pain Score | 6 months FU
  KOOS-Pain Score is referred to a subscale of pain composed by 9 items. The score range considerate is 0-100.The score uses a 5-point Likert scale and each question is assigned a score from 0 to 4, where 0 indicates "no pain" and 4 "severe level of pain".

SECONDARY OUTCOMES:
KOOS Score | baseline, 1 month, 3 months, 6 and 12 months follow-up
  KOOS SCORE consists of 5 subscales and covers: pain (9 items), symptoms (7 items, two of which are related to stiffness), functions and activities of daily living (17 items), physical function, sports and leisure activities (5 items) and quality of life in relation to the knee (4 items).
  Each question is scored from 0 to 4, where 0 indicates "no difficulty" and 4 "severe difficulty. Score range 0-100 for each subscale
IKDC-Subjective Score | baseline, 1 month, 3 months, 6 and 12 months follow-up
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathologies. All questions examines 3 categories: symptoms, sports activity, and knee function.
Visual Analogue Scale (VAS) | baseline, 1 month, 3 months, 6 and 12 months follow-up
  VAS is a visual analogue scale consisting of a range scale (10 cm length), the ends of which correspond to "no pain" and "the strongest pain imaginable".
EQ-VAS | baseline, 1 month, 3 months, 6 and 12 months follow-up
  EQ-VAS Is a visual analog scale that has a range of scores from 0 (worst imaginable health condition) to 100 (best imaginable health condition).
EQ-5D (EuroQoL) Current Health Assessment | baseline, 1 month, 3 months, 6 and 12 months follow-up
  EQ-5D is useful to evaluate the quality life of the patients
Tegner Activity Level Scale | baseline, 1 month, 3 months, 6 and 12 months follow-up
  Tegner activity level scale allows to know the level of physical activity carried out by the patients. All patients will indicate the type of sporting activity performed and its frequency.
Objective parameters- Range of Motion | baseline, 1 month, 3 months, 6 and 12 months follow-up
  Evaluation of the Range of Motion for comparative analysis.
Patient Acceptable Symptom State (PASS) | baseline, 1 month, 3 months, 6 and 12 months follow-up
  A tool to assess patient satisfaction in consideration of their current degree of pain, function, and daily activity. Patients can express if their state of health will be satisfying, answering "yes" or "no.
Objective parameters - Circumferences | baseline, 1 month, 3 months, 6 and 12 months follow-up
  Bilateral trans- and supra- patellar circumferences measurement for comparative analysis

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Di Martino, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Martino A, Di Matteo B, Papio T, Tentoni F, Selleri F, Cenacchi A, Kon E, Filardo G. Platelet-Rich Plasma Versus Hyaluronic Acid Injections for the Treatment of Knee Osteoarthritis: Results at 5 Years of a Double-Blind, Randomized Controlled Trial. Am J Sports Med. 2019 Feb;47(2):347-354. doi: 10.1177/0363546518814532. Epub 2018 Dec 13. PMID 30545242
- [Background] Filardo G, Kon E, Pereira Ruiz MT, Vaccaro F, Guitaldi R, Di Martino A, Cenacchi A, Fornasari PM, Marcacci M. Platelet-rich plasma intra-articular injections for cartilage degeneration and osteoarthritis: single- versus double-spinning approach. Knee Surg Sports Traumatol Arthrosc. 2012 Oct;20(10):2082-91. doi: 10.1007/s00167-011-1837-x. Epub 2011 Dec 28. PMID 22203046
- [Background] Braun HJ, Kim HJ, Chu CR, Dragoo JL. The effect of platelet-rich plasma formulations and blood products on human synoviocytes: implications for intra-articular injury and therapy. Am J Sports Med. 2014 May;42(5):1204-10. doi: 10.1177/0363546514525593. Epub 2014 Mar 14. PMID 24634448
- [Background] Cavallo C, Filardo G, Mariani E, Kon E, Marcacci M, Pereira Ruiz MT, Facchini A, Grigolo B. Comparison of platelet-rich plasma formulations for cartilage healing: an in vitro study. J Bone Joint Surg Am. 2014 Mar 5;96(5):423-9. doi: 10.2106/JBJS.M.00726. PMID 24599205
- [Background] Everts PA, Knape JT, Weibrich G, Schonberger JP, Hoffmann J, Overdevest EP, Box HA, van Zundert A. Platelet-rich plasma and platelet gel: a review. J Extra Corpor Technol. 2006 Jun;38(2):174-87. PMID 16921694